CLINICAL TRIAL: NCT00077389
Title: Intensified Pre-Operative Chemotherapy And Radical Surgery For High Risk Hepatoblastoma
Brief Title: Intensive Neoadjuvant Chemotherapy in Treating Young Patients Undergoing Surgical Resection for High-Risk Hepatoblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000350221; SIOP-SIOPEL-4; EU-20336; CCLG-LT-2004-09
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2009-12

CONDITIONS: Liver Cancer
Keywords: childhood hepatoblastoma; stage IV childhood liver cancer
MeSH Terms: conditions — Liver Neoplasms; Hepatoblastoma | interventions — Carboplatin; Cisplatin; Doxorubicin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: doxorubicin hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well neoadjuvant chemotherapy works in treating young patients who are undergoing surgical resection for high-risk hepatoblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy and short-term toxicity of intensified neoadjuvant chemotherapy in children with high-risk hepatoblastoma undergoing surgical resection.
* Increase the rate of complete surgical resection in these patients by fully implementing liver transplantation as a valid treatment option for tumor removal when partial liver resection or other surgical options remain unfeasible even after extensive preoperative chemotherapy.
* Determine, prospectively, the role of this regimen in rendering unresectable tumors resectable in these patients.
* Determine the accuracy of initial imaging in predicting the surgical options (after treatment with this regimen) for patients presenting with unresectable disease.

Secondary

* Determine the overall survival and event-free survival of patients treated with this regimen (with an acceptable overall toxicity).
* Determine the toxicity of this regimen in these patients.
* Determine the response rate in patients treated with this regimen.
* Determine whether response to this regimen, defined by the modified RECIST criteria, can be used for better monitoring of response in these patients.
* Determine whether a fall in alpha-fetoprotein during this neoadjuvant regimen can be used as a prognostic factor in these patients.
* Determine, prospectively, radiological, surgical, and pathological characteristics of the tumor that might identify possible novel factors that might influence treatment choice and outcome in these patients.

OUTLINE: This is an open-label, multicenter study.

* Intensified neoadjuvant chemotherapy: Patients receive cisplatin IV over 24 hours on days 1, 8, 15, 29, 36, 43, 57, and 64; and doxorubicin IV over 1 hour OR over 24 hours on days 8, 9, 36, 37, 57, and 58. Patients determined to have resectable disease proceed to surgery.

Patients determined to have unresectable disease after neoadjuvant chemotherapy receive additional neoadjuvant chemotherapy comprising carboplatin IV over 1 hour on days 1 and 22 and doxorubicin IV over 1 hour OR over 24 hours on days 1, 2, 3, 22, 23, and 24.

Treatment continues in the absence of unacceptable toxicity.

* Surgery: Patients determined to have resectable disease undergo complete resection and possibly liver transplantation.
* Adjuvant chemotherapy*: Patients who undergo complete surgical resection receive carboplatin IV over 1 hour on day 1 and doxorubicin IV over 1 hour OR over 24 hours on days 1 and 2. Treatment repeats every 3 weeks for a total of 3 courses.

NOTE: *Patients who received additional neoadjuvant chemotherapy for unresectable disease do not receive adjuvant chemotherapy.

Patients are followed every 2-3 months for 2 years, every 3 months for 1 year, and then every 6 months for 2 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 23-57 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatoblastoma
* High-risk disease, meeting criteria for at least 1 of the following:

  * Tumor involving all 4 hepatic sections
  * Evidence of abdominal extrahepatic disease
  * Presence of metastases
  * Alpha-fetoprotein < 100 ng/mL at diagnosis
* Must have had a prior diagnostic biopsy within the past 15 days
* No recurrent disease

PATIENT CHARACTERISTICS:

Age

* Under 18

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* AST and/or ALT ≤ 3 times normal

Renal

* Glomerular filtration rate ≥ 60 mL/min

Cardiovascular

* Shortening fraction ≥ 29% OR
* Ejection fraction ≥ 40%

Other

* Not pregnant
* Negative pregnancy test
* No pre-existing clinically relevant bilateral hearing loss
* No other condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for hepatoblastoma

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Estimated)
Dates: Start 2004-01

PRIMARY OUTCOMES:
Rate of complete remission after completion of study therapy

SECONDARY OUTCOMES:
Complete resection rate
Response rate to preoperative chemotherapy
Rate of grade 2 cardiac and renal, grade 3 otological, and grade 4 nonhematological toxicity as assessed during and after completion of study therapy
Overall survival
Event-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Childs, Study Chair — Children's Cancer and Leukaemia Group
Locations (24):
- Institut Gustave Roussy, Villejuif, France
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Emma Kinderziekenhuis, Amsterdam, Netherlands
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Children's Cancer and Leukaemia Group, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Derived] Zsiros J, Brugieres L, Brock P, Roebuck D, Maibach R, Zimmermann A, Childs M, Pariente D, Laithier V, Otte JB, Branchereau S, Aronson D, Rangaswami A, Ronghe M, Casanova M, Sullivan M, Morland B, Czauderna P, Perilongo G; International Childhood Liver Tumours Strategy Group (SIOPEL). Dose-dense cisplatin-based chemotherapy and surgery for children with high-risk hepatoblastoma (SIOPEL-4): a prospective, single-arm, feasibility study. Lancet Oncol. 2013 Aug;14(9):834-42. doi: 10.1016/S1470-2045(13)70272-9. Epub 2013 Jul 4. PMID 23831416
- [Derived] Weeda VB, Murawski M, McCabe AJ, Maibach R, Brugieres L, Roebuck D, Fabre M, Zimmermann A, Otte JB, Sullivan M, Perilongo G, Childs M, Brock P, Zsiros J, Plaschkes J, Czauderna P, Aronson DC. Fibrolamellar variant of hepatocellular carcinoma does not have a better survival than conventional hepatocellular carcinoma--results and treatment recommendations from the Childhood Liver Tumour Strategy Group (SIOPEL) experience. Eur J Cancer. 2013 Aug;49(12):2698-704. doi: 10.1016/j.ejca.2013.04.012. Epub 2013 May 15. PMID 23683550